CLINICAL TRIAL: NCT06248177
Title: Effect of a Probiotic Consumption on Gastrointestinal Symptoms in Adults Men and Women (FLORABIOTIC REFUERZO).
Brief Title: Probiotic Effect on Gastrointestinal Symptoms (FLORABIOTIC REFUERZO).
Acronym: FLORABIOTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023.199
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-01

CONDITIONS: Probiotic; Gastrointestinal Symptoms; Microbiota
Keywords: Microbiota; Gastrointestinal symptoms; Probiotic; Humans; Crossover
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomised, double blinded, crossover intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The products (experimental and placebo), will be produced by an external producer, who will save the codes. None of the researchers involved in the study development or analyses will know the association until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): 6 weeks daily consumption of one probiotic capsule + 4 weeks wash-out period+ 6 weeks daily consumption of one placebo capsule
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Placebo
- Group 2 (Active Comparator): 6 weeks daily consumption of one placebo capsule + 4 weeks wash-out period+ 6 weeks daily consumption of one probiotic capsule
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic capsules
Dietary Supplement: Placebo — Placebo capsules

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effect on the microbiota and the reduction in the number and/or intensity of symptoms of gastrointestinal discomfort of consuming a probiotic or placebo for 6 weeks in adult women and men.

The main questions to answer are:

1. To study changes in the alpha diversity of the microbiota.
2. To evaluate changes in the salivary cortisol.

For this purpose, a randomized, double blind crossover study has been designed.

Target sample size is 30 subjects.

Participants will be allocated in two groups for 16 weeks (6 weeks consuming one of the products + 4 weeks wash-out period + 6 weeks consuming the other product).

* Group 1 (n=15): 6 weeks daily consumption of one probiotic capsule + 4 weeks wash-out period+ 6 weeks daily consumption of one placebo capsule.
* Group 2 (n=15): 6 weeks daily consumption of one placebo capsule + 4 weeks wash-out period+ 6 weeks daily consumption of one probiotic capsule.

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study will be interviewed by phone to verify that they meet the main inclusion criteria. Volunteers who meet the main inclusion criteria will be invited to an information and screening visit to resolve any doubts. Volunteers who agree to participate in the study will sign the informed consent and will be randomly allocated to one of the two arms of the study and will be provided with any required material.

During the intervention, volunteers will attend 4 visits distributed in two phases of 6 weeks separated by 4 weeks of wash-out period. At the beginning and at the end of each phase there will be a clinical visit. In all visits anthropometric and body composition measurements, stool and saliva samples, as well as data about dietary and physical activity will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes aged between 18 and 65 years old.
* Volunteers with a body mass index between 18.5 and 30 kg/m2.
* Present some type of discomfort/discomfort at gastrointestinal levels without having a specific diagnosis.The gastrointestinal symptoms rating scale will be used to more objectively detect these symptoms. A score between 3 and 5 in any of the symptoms will be an inclusion criterion.
* Present a stable weight (+/- 3 kg) in the last three months prior to the start of the study.
* Subjects must be able to understand and be willing to sign the informed consent, and must comply with all study procedures and requirements.

Exclusion Criteria:

* Subjects with relevant functional or structural anomalies of the digestive system, such as malformations, angiodysplasias, active peptic ulcers, chronic inflammatory or malabsorption diseases, hiatal hernia, reflux with medication, helicobacter pylori, celiac disease and other diagnosed intolerances, etc.
* Subjects with surgical interventions with permanent consequences in the digestive system (for example, gastroduodenostomy).
* Subjects following treatments that alter gastrointestinal function, either chronically or occasionally.
* Subjects who are being treated with antibiotics (in order to participate, they do not have to have taken antibiotics during the two months prior to the baseline visit).
* Subjects with any type of cancer or undergoing treatment for it, or with less than 5 years since its eradication.
* Subjects with any liver disease (may participate with non-alcoholic fatty liver disease).
* Subjects with allergy to any component of the product under study.
* Subjects with a high alcohol intake, more than 14 units/day (women) and 20 units/day (men).
* Pregnant or breastfeeding women.
* Subjects who present some type of cognitive and/or psychological impediment.
* Subjects in whom poor collaboration is expected or with difficulties in following the study procedures.
* Subjects who work with shift changes that include nights.
* Subjects who follow any type of supplementation that interferes with the study (example: other probiotics).
* Subjects who are immersed in a significant lifestyle change.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota | Clinical Investigation Days 1, 2, 3 and 4.
  Fecal microbiota of participants will be analyzed by bacterial 16S gene sequencing technology.

SECONDARY OUTCOMES:
Salivary cortisol | Clinical Investigation Days 1, 2, 3 and 4 (at wake up in the morning, and at the same time in each Clinical investigation days).
  Cortisol levels will be taken by Salivette®- Cortisol kit and analyzed by electrochemiluminescence immunoassay and reported in ug/dL.
Body weight | Clinical Investigation Days 1, 2, 3 and 4
  Weight of participants will be measured by bioimpedance and reported in kg
Height | Clinical Investigation Day 1
  Height of participants will be measured by stadiometer and reported in m.
Body mass index | Clinical Investigation Days 1, 2, 3 and 4
  Body mass index will be calculated as follows: weight (kg)/ height (cm)2.
Body fat percentage | Clinical Investigation Days 1, 2, 3 and 4
  Body fat of participants will be analyzed by bioimpedance and reported in percentage and kilograms.
Body muscle mass | Clinical Investigation Days 1, 2, 3 and 4
  Body muscle mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body lean mass | Clinical Investigation Days 1, 2, 3 and 4
  Body lean mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body water mass | Clinical Investigation Days 1, 2, 3 and 4
  Body water mass of participants will be analyzed by bioimpedance and reported in kilograms.
Body bone mass | Clinical Investigation Days 1, 2, 3 and 4
  Body bone mass of participants will be analyzed by bioimpedance and reported in kilograms.
Gastrointestinal symptoms | Clinical Investigation Days 1, 2, 3 and 4
  Gastrointestinal symptoms will be registrated through 15 items likert questionnaire; gastrointestinal symptoms rating scale questionnaire.
Dietary intake | Clinical Investigation Days 1, 2, 3 and 4
  Dietary intake will be analysed by food frequency questionnaire.
Physical activity | Clinical Investigation Days 1, 2, 3 and 4
  Physical activity will be evaluated by the reduced version of the International Physical Activity Questionnaire (IPAQ).
Adherence to capsule consumption | Clinical Investigation Days 1, 2, 3 and 4
  Adherence will be assessed using the capsule consumption record form.

CONTACTS AND LOCATIONS:
Overall Officials: Fermín I Milagro Yoldi, PhD, Principal Investigator — University of Navarra; Idoia Ibero-Baraibar, PhD, Study Chair — University of Navarra; Carlos González-Navarro, PhD, Study Chair — University of Navarra; Santiago Navas-Carretero, PhD, Study Chair — University of Navarra; Gabriela Arias, Study Chair — University of Navarra; Roncesvalles Garayoa, PhD, Study Chair — University of Navarra; María Goñi, Study Chair — University of Navarra; Salomé Pérez, Study Chair — University of Navarra
Locations (1):
- Centre for Nutrition Research, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No